CLINICAL TRIAL: NCT00143507
Title: Effects of Ivabradine on Cardiovascular Events in Patients With Stable Coronary Artery Disease and Left Ventricular Systolic Dysfunction. A Three-year Randomised Double-blind Placebo-controlled International Multicentre Study.
Brief Title: The BEAUTIFUL Study: Effects of Ivabradine in Patients With Stable Coronary Artery Disease and Left Ventricular Systolic Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-16257-056
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Coronary Disease; Ventricular Dysfunction, Left
MeSH Terms: conditions — Coronary Disease; Ventricular Dysfunction, Left | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ivabradine (Experimental)
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine
  Arms: Ivabradine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to test whether ivabradine is able to reduce cardiovascular events when given to patients with coronary artery disease and impaired heart function.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Left ventricular systolic dysfunction
* Sinus rhythm: heart rate (HR) >= 60 beats per minute (bpm)

Exclusion Criteria:

* Unstable cardiovascular condition
* Severe congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10917 (Actual)
Dates: Start 2004-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Fox, MD, Study Chair — Royal Brompton National Heart and Lung Hospital
Locations (1):
- Royal Brompton National Heart and Lung Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were men and women, with documented history of coronary artery disease, associated with left ventricular systolic dysfunction. Angina and/or heart failure symptoms should have been stable for ≥ 3 months, with optimal conventional cardiovascular medication on appropriate stable doses for at least 1 month.
Pre-assignment Details: Following a run-in period of two weeks during which no study treatment was dispensed, the participants were randomised to receive ivabradine or placebo in addition to their usual cardiovascular treatment in double-blind treatment period.
Groups:
- Ivabradine: Patients received ivabradine at starting dose of 5 mg twice daily, with a target dose, if HR tolerance criteria were met after two weeks (at the D15 visit), of 7.5 mg twice daily.
- Placebo: Patients received placebo twice daily.
Period: Overall Study
Arm/Group | Ivabradine | Placebo
Started | 5479 | 5438
Completed | 4792 | 4786
Not Completed | 687 | 652
Not completed — Death | 572 | 547
Not completed — Withdrawal by Subject | 114 | 102
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawn by sponsor's decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine | Placebo | Total
Number analyzed (Participants) | 5479 | 5438 | 10917
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.5) | 65 (8.4) | 65.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 939 | 931 | 1870
  Male | 4540 | 4507 | 9047
Beta-blocker intake [Number; unit: participants]
  Yes | 4749 | 4738 | 9487
  No | 730 | 700 | 1430

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Endpoint
Description: First event among cardiovascular death, hospitalisation for acute myocardial infarction (fatal or not), or hospitalisation for new onset or worsening heart failure (fatal or not).
Time Frame: From the date of randomisation to the date of the first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 844 | 832
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.945, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.91 to 1.10] — Estimate of the hazard ratio between treatment groups based on an adjusted Cox proportional hazards model with beta-blocker intake as a covariate. P-value: Log-rank test stratified on beta-blocker intake factor

2. Secondary Outcome: Cardiovascular Death
Description: Cardiovascular death including sudden death of unknown cause
Time Frame: From the date of randomisation to death, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 469 | 435
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.316, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.94 to 1.22] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Hospitalisation for Acute Myocardial Infarction
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 3 years.
Measure: Number; unit: Participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
Participants | 199 | 226
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.159, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.06] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Hospitalisation for New Onset or Worsening Heart Failure
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 426 | 427
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.850, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.13] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: All-cause of Mortality
Time Frame: From the date of randomisation to death, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 572 | 547
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.547, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.92 to 1.16] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Coronary Artery Disease Death
Description: Death due to heart failure, acute myocardial infarction or cardiac procedure
Time Frame: From the date of randomisation to death, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 136 | 151
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.331, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.71 to 1.12] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Hospitalisation for Coronary Revascularisation
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 155 | 186
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.078, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.67 to 1.02] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Hospitalisation for Unstable Angina
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 114 | 105
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.583, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.83 to 1.40] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Hospitalisation for Acute Coronary Syndrome (Unstable Angina or Acute Myocardial Infarction)
Time Frame: From the date of randomisation to the date of first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 303 | 317
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.501, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.81 to 1.11] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Hospitalisation for Acute Coronary Syndrome, or Coronary Revascularisation
Time Frame: From the date of randomisation to the date of first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 364 | 401
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.141, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.78 to 1.04] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Hospitalisation for Acute Coronary Syndrome, New Onset or Worsening Heart Failure or Coronary Revascularisation
Time Frame: From the date of randomisation to the date of first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 681 | 704
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.411, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.86 to 1.06] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Cardiovascular Death, or Hospitalisation for New Onset or Worsening Heart Failure
Time Frame: From the date of randomisation to the date of first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 757 | 723
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.484, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.94 to 1.15] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Cardiovascular Death, or Hospitalisation for Acute Myocardial Infarction
Time Frame: From the date of randomisation to the date of the first occurrence of the first event, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 5479 | 5438
participants | 606 | 593
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.835, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.90 to 1.13] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From randomization to death, up to 3 years
Description: The Randomised Set consisted of 10 917 patients (5479 patients in the ivabradine group and 5438 patients in the placebo group). The Safety Set consisted of 10 907 patients: 10 randomised patients were excluded from the Safety Set because they did not take any study drug (2 patients in the ivabradine group and 8 patients in the placebo group).
Arm/Group | Ivabradine | Placebo
Serious Adverse Events (participants affected / at risk) | 1625/5477 | 1770/5430
Other Adverse Events (participants affected / at risk) | 2570/5477 | 2221/5430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=5477) | Placebo (N=5430)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 9 (11)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 16 (18) | 21 (22)
Acute left ventricular failure (Cardiac disorders) | 19 (22) | 18 (18)
Acute myocardial infarction (Cardiac disorders) | 82 (85) | 88 (96)
Angina pectoris (Cardiac disorders) | 37 (38) | 66 (73)
Angina unstable (Cardiac disorders) | 153 (182) | 197 (223)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 127 (145) | 134 (162)
Atrial flutter (Cardiac disorders) | 35 (38) | 28 (30)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
Atrioventricular block complete (Cardiac disorders) | 10 (10) | 12 (12)
Atrioventricular block second degree (Cardiac disorders) | 8 (8) | 7 (7)
Bradycardia (Cardiac disorders) | 22 (22) | 6 (6)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac asthma (Cardiac disorders) | 5 (5) | 4 (5)
Cardiac failure (Cardiac disorders) | 405 (517) | 438 (584)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 7 (7)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 13 (15) | 19 (19)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 6 (6) | 8 (8)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 4 (4)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 67 (71) | 81 (83)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 8 (8) | 2 (2)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 2 (2) | 3 (3)
Sinus arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 4 (4) | 2 (2)
Ventricular bigeminy (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 8 (8) | 7 (7)
Ventricular fibrillation (Cardiac disorders) | 16 (16) | 13 (13)
Ventricular tachycardia (Cardiac disorders) | 28 (28) | 53 (58)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital intestinal malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Epidermal naevus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 6 (6)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular neuronitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypercorticoidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyrotoxicosis (Endocrine disorders) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 8 (9) | 6 (6)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 1 (1)
Exophthalmos endocrine (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 2 (2)
Retinal artery occlusion (Eye disorders) | 1 (1) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 7 (7) | 5 (5)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 14 (14) | 22 (22)
Inguinal hernia gangrenous (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric occlusion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal stenosis acquired (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pancreatitis due to biliary obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perirectal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Application site reaction (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 15 (15) | 21 (22)
Death (General disorders) | 37 (37) | 26 (26)
Difficulty in walking (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 8 (8)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Sudden death (General disorders) | 204 (204) | 185 (185)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 0 (0)
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 6 (6)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 6 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 15 (15) | 13 (13)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytolytic hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic oedema (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 5 (5)
Appendicitis (Infections and infestations) | 3 (3) | 3 (3)
Aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 3 (9)
Bronchitis acute (Infections and infestations) | 10 (10) | 8 (8)
Bronchitis acute viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis chronic (Infections and infestations) | 5 (5) | 10 (11)
Bronchopneumonia (Infections and infestations) | 6 (6) | 4 (4)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dental caries (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 3 (3) | 0 (0)
Diphyllobothriasis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 2 (2) | 6 (6)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 10 (10)
Gastroenteritis Norwalk virus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 2 (2) | 4 (4)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 3 (3) | 10 (10)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 71 (75) | 64 (72)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Postoperative infection (Infections and infestations) | 0 (0) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 2 (2) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 5 (7)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Superinfection lung (Infections and infestations) | 2 (2) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Urosepsis (Infections and infestations) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 4 (4)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angiogram (Investigations) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 26 (26) | 28 (29)
Biopsy lung (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Cardiovascular evaluation (Investigations) | 3 (3) | 7 (7)
Catheterisation cardiac (Investigations) | 0 (0) | 2 (2)
Colonoscopy (Investigations) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 7 (7) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Investigation (Investigations) | 4 (4) | 4 (5)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Scan myocardial perfusion (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Transplant evaluation (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 26 (27) | 25 (26)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (9)
Lordosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Monoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyserositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell carcinoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Gastric cancer stage IV with metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Laryngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 11 (11)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 10 (10)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Rectosigmoid cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery atheroma (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 7 (7) | 3 (3)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atherosclerosis (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 8 (8) | 11 (11)
Cerebral ischaemia (Nervous system disorders) | 4 (4) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 38 (38) | 35 (36)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 4 (6) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 5 (5)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Facial palsy (Nervous system disorders) | 1 (1) | 1 (2)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 37 (37) | 41 (43)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 2 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 1 (1) | 5 (5)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 19 (21) | 19 (19)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 6 (6)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 18 (18) | 26 (26)
Vertebrobasilar insufficiency (Nervous system disorders) | 4 (4) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (4)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Pathological gambling (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bilateral hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 14 (14) | 5 (5)
Renal failure chronic (Renal and urinary disorders) | 4 (4) | 4 (4)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (4)
Renal insufficiency (Renal and urinary disorders) | 13 (13) | 14 (15)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 11 (11)
Hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 21 (28)
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Maxillary sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemosiderosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Diabetic gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pyoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arrhythmia prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 2 (2) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Arterial therapeutic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac aneurysm repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Cardiac operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 7 (7) | 3 (3)
Cardiac pacemaker revision (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 2 (2) | 3 (4)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 2 (2) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract extraction (Surgical and medical procedures) | 4 (4) | 2 (3)
Catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 12 (12) | 19 (19)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Coronary artery surgery (Surgical and medical procedures) | 13 (13) | 14 (14)
Coronary revascularisation (Surgical and medical procedures) | 3 (3) | 4 (4)
Diabetes mellitus management (Surgical and medical procedures) | 2 (2) | 1 (1)
Finger amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gingival operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 3 (3)
Implantable defibrillator insertion (Surgical and medical procedures) | 12 (12) | 15 (15)
Incisional hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 2 (2) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 3 (3) | 3 (3)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 2 (2)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Orchidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Penile prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Radioactive iodine therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal revascularisation surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Scar excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Thromboendarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1)
Transurethral microwave therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Varicose veins ligation (Surgical and medical procedures) | 0 (0) | 1 (1)
Vasodilation procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Wart excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 4 (4)
Aortic aneurysm rupture (Vascular disorders) | 3 (3) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial embolism limb (Vascular disorders) | 0 (0) | 4 (4)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 5 (6) | 1 (1)
Arteriopathic disease (Vascular disorders) | 0 (0) | 1 (1)
Atherosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Atherosclerosis obliterans (Vascular disorders) | 1 (1) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 16 (17) | 12 (12)
Circulatory collapse (Vascular disorders) | 1 (1) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 3 (4) | 5 (5)
Diabetic peripheral angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 2 (2) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 2 (2) | 3 (3)
Gangrene (Vascular disorders) | 6 (6) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 11 (11) | 9 (9)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 5 (5)
Iliac artery stenosis (Vascular disorders) | 2 (2) | 0 (0)
Iliac artery thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Iliac vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 5 (5) | 4 (4)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 4 (5)
Peripheral occlusive disease (Vascular disorders) | 17 (17) | 28 (30)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 2 (2) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=5477) | Placebo (N=5430)
Anaemia (Blood and lymphatic system disorders) | 61 (62) | 60 (61)
Angina pectoris (Cardiac disorders) | 100 (108) | 98 (110)
Atrial fibrillation (Cardiac disorders) | 172 (203) | 148 (167)
Bradycardia (Cardiac disorders) | 185 (189) | 50 (51)
Cardiac failure (Cardiac disorders) | 176 (198) | 188 (210)
Ventricular extrasystoles (Cardiac disorders) | 99 (102) | 95 (100)
Phosphenes (Eye disorders) | 206 (219) | 46 (49)
Chest pain (General disorders) | 47 (50) | 59 (67)
Fatigue (General disorders) | 59 (62) | 56 (60)
Oedema peripheral (General disorders) | 41 (44) | 56 (56)
Bronchitis (Infections and infestations) | 71 (83) | 80 (100)
Bronchitis acute (Infections and infestations) | 49 (53) | 61 (64)
Influenza (Infections and infestations) | 65 (74) | 73 (78)
Nasopharyngitis (Infections and infestations) | 84 (89) | 87 (98)
Pneumonia (Infections and infestations) | 56 (58) | 52 (57)
Blood cholesterol increased (Investigations) | 56 (57) | 75 (77)
Blood creatinine increased (Investigations) | 57 (61) | 53 (56)
Blood triglycerides increased (Investigations) | 59 (59) | 62 (62)
Heart rate decreased (Investigations) | 164 (164) | 34 (36)
Diabetes mellitus (Metabolism and nutrition disorders) | 68 (68) | 54 (55)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 150 (155) | 171 (192)
Gout (Metabolism and nutrition disorders) | 44 (49) | 57 (63)
Hyperkalaemia (Metabolism and nutrition disorders) | 60 (66) | 64 (66)
Dizziness (Nervous system disorders) | 103 (109) | 81 (85)
Headache (Nervous system disorders) | 55 (60) | 53 (60)
Renal insufficiency (Renal and urinary disorders) | 56 (60) | 61 (62)
Blood pressure inadequately controlled (Vascular disorders) | 181 (203) | 177 (191)
Hypotension (Vascular disorders) | 46 (50) | 70 (72)

LIMITATIONS AND CAVEATS:
The section Other Adverse Events (Not including serious) has been completed by the sponsor to include only the Non Serious Adverse Events emergent on treatment during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publication and/or communication related to the study results and can require changes. In case of a patent application, the sponsor can delay its authorization for publication or communication of the study results until the date of international registration of the patent.